CLINICAL TRIAL: NCT03079908
Title: Comparison of the da Vinci Skills Simulator and the LapSim Laparoscopy Simulator for Conventional Laparoscopic Skills Improvement: a Prospective, Randomized Trial
Brief Title: Comparison of da Vinci Simulator vs LapSim Simulator
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough resources to start the study
Sponsor: Klinik für Allgemein- und Viszeralchirurgie, Department Chirurgie, Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Pouya Iranmanesh, Oberarzt (Senior Resident), Dr. med (MD), Klinik für Allgemein- und Viszeralchirurgie, Department Chirurgie, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Simulator study
Record Dates: First submitted 2017-02-23; First posted 2017-03-15 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Laparoscopy Training; Robotic Surgery Training
Keywords: Laparoscopy; Surgery; Training; Virtual reality; Simulation; Robotic Surgery; Da Vinci

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Da Vinci Skills Simulator® (Experimental): Participants in this group will undergo robotic virtual reality surgical simulator training (Da Vinci Mimics) and will subsequently be evaluated on a dry lab laparoscopic box
  Interventions: Other: da Vinci Skills Simulator®
- LapSim® (Active Comparator): Participants in this group will undergo laparoscopic virtual reality surgical simulator Training (LapSim) and will subsequently be evaluated on a dry lab laparoscopic box
  Interventions: Other: LapSim®
- Dry lab box laparoscopic training (Placebo Comparator): Participants in this group will undergo dry lab box laparoscopic training only
  Interventions: Other: Dry lab box laparoscopic training

INTERVENTIONS:
Other: da Vinci Skills Simulator® — Initial robotic virtual reality surgical simulator Training (da Vinci Skills Simulator ® System), then laparoscopic dry box evaluation
  Arms: Da Vinci Skills Simulator®
Other: LapSim® — Initial laparoscopic virtual reality surgical simulator training (LapSim ® System), then laparoscopic dry box evaluation
  Arms: LapSim®
Other: Dry lab box laparoscopic training — No initial simulator training. Dry lab box laparoscopic Training only.
  Arms: Dry lab box laparoscopic training

SUMMARY:
Virtual reality surgical simulators (VRSS) are gaining popularity for general surgery training, both for conventional laparoscopic and robotically-assisted surgery. Although numerous studies have analysed the impact of VRSS training on surgical skills, there is a lack of data regarding the comparison of robotic VRSS (RVRSS) and laparoscopic VRSS (LVRSS) training on conventional laparoscopic skills among subjects with no prior surgical experience. The hypothesis of the present study is that RVRSS could improve conventional laparoscopic skills as much as laparoscopic LVRSS among naïve subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy medical students aged 20 to 30 years old

Exclusion Criteria:

* No prior surgical, laparoscopic or robotic experience
* No previously known severe learning disability or mental deficiency
* No handicap limiting the usage of one or both upper limb(s)

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Exercises times | Within 1 day after randomization / data will be presented after completion of the study (an average of 9 months)
  Time to realize each training exercise as well as the final evaluation exercise

SECONDARY OUTCOMES:
Objects drops | Within 1 day after randomization / data will be presented after completion of the study (an average of 9 months)
  Number of time objects were unwillingly dropped during each training exercise as well as the final evaluation exercise
Objects out of view | Within 1 day after randomization / data will be presented after completion of the study (an average of 9 months)
  Number of times one or both instruments or objects used for the exercises were out of the viewing field during each training exercise as well as the final evaluation exercise
Instruments collisions | Within 1 day after randomization / data will be presented after completion of the study (an average of 9 months)
  Number of collisions between the different instruments used to perform each training exercise as well as the final evaluation exercise

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Scheiwiller, MD, Study Director — Luzerner Kantonsspital Luzern, Switzerland
Locations (1):
- Luzern Kantonsspital Luzern, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No